CLINICAL TRIAL: NCT03338933
Title: Neurobiology of Alcohol and Nicotine Co-Addiction
Acronym: NAUD
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: NURA-002-17S; 17321 (Other: Oregon Health and Science University)
Record Dates: First submitted 2017-11-06; First posted 2017-11-09 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Use Disorder; Nicotine Use Disorder
MeSH Terms: conditions — Alcoholism; Tobacco Use Disorder | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cheek swab Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Control Group: No history of addiction to any substance or gambling. Less than 20 lifetime cigarettes or equivalent.
  Interventions: Behavioral: magnetic resonance imaging (MRI)
- Nicotine Group: Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-V) criteria for Nicotine Use Disorder. Current smoker, at least 10 cigarettes per day. No history of addiction to any other substance
  Interventions: Behavioral: magnetic resonance imaging (MRI)
- Nicotine and Alcohol Group: DSM-V criteria for Nicotine Use Disorder and Alcohol Use Disorder. At least 8 heavy drinking episodes in the past month. Current smoker. Alcohol free from 2 to 4 weeks. No history of addiction to other substances or gambling.
  Interventions: Behavioral: magnetic resonance imaging (MRI)
- Alcohol Group: DSM-V criteria for Alcohol use Disorder. At least 8 heavy drinking episodes in the past month. Abstinent for at least 2 weeks and no more than 4 weeks. Less than 20 lifetime cigarettes or equivalent. No history of addiction to any other substances or gambling.
  Interventions: Behavioral: magnetic resonance imaging (MRI)

INTERVENTIONS:
Behavioral: magnetic resonance imaging (MRI) — All subjects will undergo a baseline MRI and subjects in both alcohol groups (alcohol use disorder and combined alcohol and nicotine use disorder) will undergo a followup MRI 3 months after baseline.

SUMMARY:
This proposal addresses the critical absence of information about the neurobiology of recovery from Alcohol Use Disorder (AUD) in alcohol and nicotine users.

DETAILED DESCRIPTION:
This proposal addresses the critical absence of information about the neurobiology of recovery from Alcohol Use Disorder (AUD) in alcohol and nicotine users. AUD and nicotine use disorder (NUD) are the most commonly abused (non-prescription) substances in the U.S. Co-addiction is particularly high in military veterans. Although nationwide estimates peg the rate of AUD/NUD co-addiction at 80%, the Substance Abuse Treatment Program (SATP) at the Veterans Affairs Portland Health Care System (VAPORHCS) finds that 90% of veterans treated for AUD also meet criteria for NUD. The investigators hypothesize that a support vector machine learning algorithm will be able to use the measures to classify subjects as AUD, NUD both or neither and that the algorithm will predict outcome (sobriety or relapse) at three months.

ELIGIBILITY:
Inclusion Criteria:

* None

Exclusion Criteria:

* None

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited from the Portland VA, Oregon Health & Science University, community substance abuse treatment programs and by advertisement.
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William F Hoffman, MD PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in a hospital setting from 2018 to 2023.
Pre-assignment Details: Of 616 phone screens conducted at the VA Portland Health Care System, 171 were eligible to participate in the study, and 109 participants signed an informed consent form. 4 participants were screened out or declined participation after consent but prior to any data collection and are not included in participant flow table. Control and Nicotine group's participation was complete after baseline measurements were collected. Alcohol groups continued to next periods.
Period: Screening Visit
Arm/Group | Control Group | Nicotine Group | Alcohol Group | Nicotine and Alcohol Group
Started | 31 | 28 | 13 | 33
Completed | 28 | 18 | 11 | 25
Not Completed | 3 | 10 | 2 | 8
Not completed — Lost to Follow-up | 1 | 3 | 1 | 4
Not completed — Screen fail after consent | 2 | 7 | 1 | 4
Period: Baseline Visit
Arm/Group | Control Group | Nicotine Group | Alcohol Group | Nicotine and Alcohol Group
Started | 28 | 18 | 11 | 25
Completed | 28 | 18 | 11 | 25
Not Completed | 0 | 0 | 0 | 0
Period: Check-In Visit (Alcohol Groups Only)
Arm/Group | Control Group | Nicotine Group | Alcohol Group | Nicotine and Alcohol Group
Started | 0 | 0 | 11 | 25
Completed | 0 | 0 | 8 | 15
Not Completed | 0 | 0 | 3 | 10
Not completed — Lost to Follow-up | 0 | 0 | 2 | 9
Not completed — Deemed no longer eligible due to changes in health | 0 | 0 | 1 | 1
Period: Follow-up Visit (Alcohol Groups Only)
Arm/Group | Control Group | Nicotine Group | Alcohol Group | Nicotine and Alcohol Group
Started | 0 | 0 | 8 | 15
Completed | 0 | 0 | 7 | 13
Not Completed | 0 | 0 | 1 | 2
Not completed — Could not complete in-person items due to COVID-19 shutdown | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Participants who screened out or were lost to follow up during the screening visit are not included in baseline analysis population reporting.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Nicotine Group | Alcohol Group | Nicotine and Alcohol Group | Total
Number analyzed (Participants) | 28 | 18 | 11 | 25 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 18 | 11 | 25 | 82
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.86 (11.4) | 38.67 (8.6) | 41.45 (6.8) | 40.88 (8.7) | 38.41 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 1 | 4 | 5 | 24
  Male | 14 | 17 | 7 | 20 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 2 | 2 | 9
  Not Hispanic or Latino | 23 | 15 | 9 | 22 | 69
  Unknown or Not Reported | 3 | 0 | 0 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 1 | 0 | 5
  Asian | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 0 | 2
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 25 | 9 | 8 | 23 | 65
  More than one race | 1 | 1 | 2 | 1 | 5
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 18 | 11 | 25 | 82

OUTCOME MEASURES:

1. Primary Outcome: Brain Activation During Functional Magnetic Resonance Imaging (fMRI) in Response to a Stress Modulated Cue Induced Craving Task (DSNBACK)
Description: The DSN-back is a cognitive task used to assess working memory and attention. Participants view a sequence of letters presented on a screen, flanked by either drug-related or neutral images, and are instructed to identify matches occurring N steps earlier. Neural activation during high working memory demand condition (2-back) relative to the low working memory condition (0-back) was investigated. Inconsistent activation patterns across regions may indicate impaired neural processing in regions critical for cognitive control, emotion regulation, and reward processing, commonly reported in substance use disorders. Values closer to 0 (no change) in regions responsible for emotion regulation and cognitive control (e.g., Amygdala, ACC) may indicate reduced task-specific engagement where drug-related processes may be dominating neural activity.
Time Frame: Baseline
Population: Participants were removed from analysis due to too much motion, performing the task incorrectly, or did not perform the task during the MRI session.
Measure: Mean (Standard Deviation); unit: Percent signal change
Arm/Group | Control Group | Nicotine Group | Alcohol Group | Nicotine and Alcohol Group
Number analyzed (Participants) | 26 | 8 | 5 | 17
Percent signal change
  Anterior Cingulate Cortex | -26.1562 (163.7528) | -45.2123 (142.7251) | 18.4989 (119.7023) | -8.8848 (93.3926)
  Amygdala | -37.6450 (101.1780) | -72.3998 (160.9536) | -36.6553 (143.9042) | -17.9994 (119.2175)
  Hippocampus | -31.8272 (106.1173) | -45.4345 (124.8141) | -69.7126 (115.1060) | -37.1105 (135.3652)
  Insula | -0.7322 (152.9914) | -73.3807 (160.7811) | 61.6090 (138.2172) | -42.4399 (146.2034)
  Medial Orbital Frontal Cortex | -35.9220 (52.9373) | -22.4666 (55.9283) | 37.5445 (95.7412) | -12.6343 (42.7803)
  Nucleus Accumbens | -56.2479 (193.2017) | -121.6585 (258.8531) | -133.8492 (123.4497) | -40.6751 (112.4257)

2. Primary Outcome: Brain Activation During Resting State MRI.
Description: This outcome measures resting-state functional connectivity (rsFC) of the striatum using seed-based analysis of resting-state fMRI data. FC values, expressed as Fisher z-transformed correlation coefficients, quantify the strength of synchronization between the striatum seed region and other brain areas. Positive values indicate synchronized activity, while negative values reflect anticorrelation. Altered rsFC of the striatum, a hub for reward processing, habit formation, and executive control, is linked to alcohol and nicotine use disorders and may indicate impaired regulation of cravings and heightened sensitivity to substance-related cues. Investigating rsFC patterns may identify biomarkers of addiction severity, predict treatment outcomes, and inform potential therapeutic targets.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: correlation coefficient
Arm/Group | Control Group | Nicotine Group | Alcohol Group | Nicotine and Alcohol Group
Number analyzed (Participants) | 25 | 10 | 5 | 8
correlation coefficient
  Anterior Cingulate Cortex (ACC) | 0.1817 (0.1460) | 0.1858 (0.1576) | 0.1729 (0.0973) | 0.1308 (0.0959)
  Amygdala | 0.1293 (0.1124) | 0.1216 (0.1148) | 0.0232 (0.0903) | 0.0930 (0.0682)
  Hippocampus | 0.0391 (0.0998) | 0.0746 (0.1068) | 0.0255 (0.0791) | 0.0348 (0.0609)
  Insula | 0.2297 (0.1390) | 0.3139 (0.1958) | 0.2134 (0.1306) | 0.2386 (0.1829)
  Medial Orbital Frontal Cortex (OFC) | 0.0469 (0.0398) | 0.0574 (0.0420) | 0.0726 (0.0456) | 0.0327 (0.0397)
  Lateral OFC | 0.0769 (0.0739) | 0.1212 (0.0826) | 0.0969 (0.0587) | 0.0770 (0.0655)
  Bilateral Middle Frontal Gyrus | -0.0501 (0.0996) | -0.0128 (0.1573) | 0.0393 (0.0580) | -0.0184 (0.0974)
  Rostral ACC | 0.1610 (0.1664) | 0.2674 (0.1721) | 0.2327 (0.1361) | 0.1293 (0.1124)
  Caudal ACC | 0.1884 (0.1459) | 0.1574 (0.1361) | 0.1598 (0.1027) | 0.1323 (0.1121)
  Bilateral Anterior Insula | 0.2561 (0.1766) | 0.3575 (0.2270) | 0.2477 (0.1456) | 0.2817 (0.1945)
  Bilateral Dorsal Anterior Insula | 0.3803 (0.2124) | 0.4823 (0.2517) | 0.3249 (0.1984) | 0.3775 (0.2760)
  Bilateral Ventral Anterior Insula | 0.1541 (0.1739) | 0.2554 (0.2228) | 0.1852 (0.1200) | 0.2039 (0.1538)
  midbrain | 0.0037 (0.1067) | 0.0390 (0.0987) | 0.0380 (0.0903) | 0.0306 (0.1308)
  Right Dorsal Lateral Prefrontal Cortex | 0.0251 (0.1323) | 0.0504 (0.1995) | 0.0074 (0.0267) | 0.1052 (0.1409)
  Sub Callosal Cortex | 0.0224 (0.0582) | 0.0673 (0.0489) | 0.1034 (0.0738) | 0.0495 (0.0533)

3. Primary Outcome: Brain Cortical Thickness Assessed During MRI
Description: This outcome measures cortical thickness (millimeters) across brain regions using structural MRI. Cortical thickness reflects the integrity of gray matter and is influenced by factors such as neurodegeneration, plasticity, and development. Reductions in cortical thickness, particularly in prefrontal and limbic regions, are associated with impaired cognitive control, emotion regulation, and decision-making in substance use disorders.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Control Group | Nicotine Group | Alcohol Group | Nicotine and Alcohol Group
Number analyzed (Participants) | 29 | 12 | 9 | 22
mm
  Left caudal anterior cingulate | 2.6111 (0.2171) | 2.5421 (0.1780) | 2.5472 (0.2005) | 2.6560 (0.5697)
  Left inferior parietal cortex | 2.4885 (0.0862) | 2.4414 (0.0675) | 2.3881 (0.0586) | 2.4132 (0.5030)
  Left rostral anterior cingulate | 2.7960 (0.1675) | 2.7058 (0.1977) | 2.7173 (0.1454) | 2.7150 (0.5749)
  Left rostral middle frontal cortex | 2.4701 (0.0898) | 2.4315 (0.0752) | 2.3740 (0.0794) | 2.4406 (0.5069)
  Left supramarginal cortex | 2.6022 (0.1315) | 2.5550 (0.0838) | 2.4669 (0.0656) | 2.5375 (0.5283)
  Right caudal anterior cingulate | 2.4662 (0.1935) | 2.4350 (0.1495) | 2.3582 (0.1392) | 2.4452 (0.5130)
  Right inferior parietal cortex | 2.5510 (0.0803) | 2.5175 (0.0953) | 2.4377 (0.0324) | 2.4774 (0.5158)
  Right rostral anterior cingulate | 2.8013 (0.1454) | 2.6618 (0.2390) | 2.6828 (0.1466) | 2.7507 (0.5852)
  Right rostral middle frontal cortex | 2.3994 (0.1024) | 2.3699 (0.0777) | 2.3103 (0.0640) | 2.3443 (0.4864)
  Right supramarginal cortex | 2.6165 (0.1221) | 2.5694 (0.0666) | 2.4713 (0.0701) | 2.5312 (0.5261)

4. Primary Outcome: Brain White Matter Integrity as Assessed by Fractional Anisotropy During MRI
Description: Fractional Anisotropy (FA) is a scalar metric derived from diffusion-weighted MRI that quantifies the degree of directional dependence (anisotropy) of water diffusion in brain white matter, with values ranging from 0 (isotropic diffusion) to 1 (maximally anisotropic diffusion). Increases in FA may reflect greater white matter organization and integrity, while decreases often indicate microstructural damage, demyelination, or axonal loss. FA measurements were averaged within predefined regions of interest (ROIs) to assess the integrity of white matter in various brain regions associated with cognitive, motor, and emotional processing. Decreased FA in tracts such as the corpus callosum or prefrontal pathways may reflect impaired communication between brain regions involved in reward processing and cognitive control in substance use disorders.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Control Group | Nicotine Group | Alcohol Group | Nicotine and Alcohol Group
Number analyzed (Participants) | 19 | 10 | 3 | 15
Unitless
  Forceps Major | 0.4167 (0.1984) | 0.3996 (0.1497) | 0.4030 (0.1900) | 0.4044 (0.1930)
  Forceps Minor | 0.3794 (0.1809) | 0.3657 (0.1374) | 0.3574 (0.1685) | 0.3589 (0.1718)
  Left Anterior Thalamic Radiation | 0.3474 (0.1653) | 0.3362 (0.1257) | 0.3356 (0.1582) | 0.3334 (0.1592)
  Right Anterior Thalamic Radiation | 0.3450 (0.1642) | 0.3337 (0.1247) | 0.3331 (0.1570) | 0.3306 (0.1578)
  Left Inferior fronto-occipital fasciculus | 0.3536 (0.1684) | 0.3388 (0.1268) | 0.3383 (0.1595) | 0.3374 (0.1614)
  Right Inferior fronto-occipital fasciculus | 0.3574 (0.1702) | 0.3436 (0.1287) | 0.3422 (0.1614) | 0.3417 (0.1632)
  Left Temporal Superior longitudinal fasciculus | 0.3535 (0.1683) | 0.3389 (0.1269) | 0.3392 (0.1600) | 0.3387 (0.1620)
  Right Temporal Superior longitudinal fasciculus | 0.3460 (0.1647) | 0.3338 (0.1251) | 0.3340 (0.1574) | 0.3330 (0.1592)
  Left Corticospinal tract | 0.3909 (0.1860) | 0.3790 (0.1418) | 0.3826 (0.1804) | 0.3800 (0.1812)
  Right Corticospinal tract | 0.3870 (0.1841) | 0.3766 (0.1407) | 0.3802 (0.1792) | 0.3780 (0.1802)
  Left cingulate gyrus | 0.3831 (0.1826) | 0.3697 (0.1385) | 0.3662 (0.1726) | 0.3652 (0.1747)
  Right cingulate gyrus | 0.3758 (0.1789) | 0.3647 (0.1364) | 0.3705 (0.1747) | 0.3662 (0.1751)
  Left Uncinate fasciculus | 0.3219 (0.1533) | 0.3136 (0.1177) | 0.3104 (0.1464) | 0.3057 (0.1463)
  Right Uncinate fasciculus | 0.3231 (0.1538) | 0.3120 (0.1172) | 0.3148 (0.1484) | 0.3073 (0.1470)
  Left Inferior longitudinal fasciculus | 0.3552 (0.1692) | 0.3388 (0.1269) | 0.3408 (0.1607) | 0.3421 (0.1636)
  Right Inferior longitudinal fasciculus | 0.3522 (0.1677) | 0.3392 (0.1272) | 0.3399 (0.1603) | 0.3393 (0.1621)
  Left Hippocampus | 0.3572 (0.1705) | 0.3464 (0.1300) | 0.3493 (0.1649) | 0.3441 (0.1645)
  Right Hippocampus | 0.3750 (0.1786) | 0.3677 (0.1377) | 0.3617 (0.1706) | 0.3635 (0.1737)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Control Group | Nicotine Group | Alcohol Group | Nicotine and Alcohol Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/28 | 0/13 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/28 | 0/13 | 0/33
Other Adverse Events (participants affected / at risk) | 0/31 | 0/28 | 0/13 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT03338933/Prot_SAP_000.pdf